CLINICAL TRIAL: NCT02492451
Title: Endometrial Injury Versus Luteal Phase Support in Intrauterine Insemination Cycles
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems in recruitment
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Selcuk Selcuk, Medical Doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zeynepkamil
Record Dates: First submitted 2015-06-18; First posted 2015-07-08 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy
Keywords: intrauterine insemination; pregnancy rate; endometrial injury
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endometrial Injury (Active Comparator): Endometrial injury in luteal phase of preceding IUI cycle
  Interventions: Other: Endometrial Injury
- Luteal Phase Support (Active Comparator): Luteal phase support with progesterone (Crinone® %8 vaginal progesterone gel) in IUI cycle Vaginal progesterone gel is administered from second day after insemination until pregnancy testing and is continued in the presence of pregnancy until the 12 weeks of pregnancy.
  Interventions: Drug: progesterone (Crinone® %8 vaginal progesterone gel)
- Control group (No Intervention): Only IUI

INTERVENTIONS:
Other: Endometrial Injury — Endometrial injury in luteal phase of preceding cycle by pipelle canula
  Arms: Endometrial Injury
Drug: progesterone (Crinone® %8 vaginal progesterone gel) — Luteal phase support with progesterone (Crinone® %8 vaginal progesterone gel) in IUI cycle Vaginal progesterone gel is administered from second day after insemination until pregnancy testing and is continued in the presence of pregnancy until the 12 weeks of pregnancy.
  Arms: Luteal Phase Support

SUMMARY:
The investigators will try to assess the effect of endometrial injury preceding the intrauterine insemination cycle on the pregnancy rates compared to cycles with luteal phase support and the control group.

DETAILED DESCRIPTION:
Group 1: Endometrial biopsy is performed on days 21-24 of the spontaneous menstrual cycle proceeding the intrauterine insemination (IUI) treatment cycle. Two small biopsies are obtained from anterior and posterior walls of the uterus.

Group 2: Vaginal progesterone gel is administered for luteal phase support from second day after insemination until pregnancy testing and is continued in the presence of pregnancy until the 12 weeks of pregnancy.

Goup 3: Patients are undergone intrauterine insemination (IUI) cycles stimulated with gonadotropin without any intervention.

The effect of endometrial injury and luteal phase progesterone support on the pregnancy rate in patients intrauterine insemination (IUI) cycles stimulated with gonadotropin will be compared in terms of biochemical pregnancy rate, clinical pregnancy rate and ongoing pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients are undergone intrauterine insemination with gonadotropin stimulation
* Bilateral patent fallopian tubes revealed by hysterosalpingography or laparoscopy
* After semen preparation for intrauterine insemination, total progressive sperm count > 5 million

Exclusion Criteria:

* endocrin or metabolic disorders,
* uterine factor,
* pelvic inflammatory disease,
* women with basal follicle-stimulating hormone (FSH) level >15 IU/mL,
* body mass index (BMI) ≥ 35 kg/m2,
* age ≥ 40 and < 18 years,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk Selcuk, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Bui BN, Lensen SF, Gibreel A, Martins WP, Torrance H, Broekmans FJ. Endometrial injury for pregnancy following sexual intercourse or intrauterine insemination. Cochrane Database Syst Rev. 2022 Oct 24;10(10):CD011424. doi: 10.1002/14651858.CD011424.pub4. PMID 36278845
- [Derived] Bui BN, Lensen SF, Gibreel A, Martins WP, Torrance H, Broekmans FJ. Endometrial injury for pregnancy following sexual intercourse or intrauterine insemination. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD011424. doi: 10.1002/14651858.CD011424.pub3. PMID 33734431

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Only intrauterine insemination
Period: Overall Study
Arm/Group | Endometrial Injury | Luteal Phase Support | Control Group
Started | 40 | 39 | 39
Completed | 40 | 39 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Injury | Luteal Phase Support | Control Group | Total
Number analyzed (Participants) | 40 | 39 | 39 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.85 (5.45) | 28.13 (4.41) | 29.95 (5.44) | 28.64 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 39 | 118
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate
Description: ongoing pregnancy rates
Time Frame: 12 weeks
Measure: Number; unit: percentage of ongoing pregnancies
Arm/Group | Endometrial Injury | Luteal Phase Support | Control Group
Number analyzed (Participants) | 40 | 39 | 39
percentage of ongoing pregnancies | 7.5 | 17.9 | 5.1

ADVERSE EVENTS:
Arm/Group | Endometrial Injury | Luteal Phase Support | Control Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes